CLINICAL TRIAL: NCT00446849
Title: A Phase IV, Multi-center, Open-label Study to Assess Clinical Recurrence Related to Compliance With Treatment With MMX Mesalamine 2.4g/Day Given Once Daily for the Maintenance of Quiescent Ulcerative Colitis (UC)
Brief Title: Strategies in Maintenance for Patients Receiving Long-term Therapy (S.I.M.P.L.E.) With MMX (Multi-Matrix System) Mesalamine for Ulcerative Colitis (UC)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD476-404
Record Dates: First submitted 2007-03-12; First posted 2007-03-13 (Estimated); Results first posted 2010-07-08 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Ulcerative Colitis
Keywords: ulcerative colitis; compliance; mesalamine; clinical study; clinical trial; clinical research; maintenance; long term; uc study; uc trial; uc research; open label; once a day; once; daily; daily dosing; simple; oral
MeSH Terms: conditions — Colitis, Ulcerative; Patient Compliance; Charcot-Marie-Tooth disease, Type 1C | interventions — Mesalamine

ARMS (1):
- MMX Mesalamine (Experimental)
  Interventions: Drug: MMX Mesalamine

INTERVENTIONS:
Drug: MMX Mesalamine — MMX™ mesalamine 2.4g/day to 4.8g/day once-daily (QD) (two to four 1.2g tablets MMX™ mesalamine, dosed QD,respectively).
  Other Names: Lialda

SUMMARY:
To evaluate the percentage of subjects with clinical recurrence of UC at 6 months using MMX mesalamine once daily.

ELIGIBILITY:
Inclusion Criteria - Acute Phase:

1. Male and female subjects aged at least 18 years with active mild to moderate UC may enter the Acute Phase of the study.
2. Must have a previous diagnosis of UC confirmed by histology and endoscopy or radiology.
3. Males or non-pregnant, non-lactating FOCP who have a negative serum pregnancy test prior to entering the study and who are using adequate forms of contraception for the duration of the study.
4. General medical assessment must be satisfactory and there must not be clinically significant and relevant abnormalities.
5. Subject must have had >2 acute episodes of UC (a documented episode of increased bowel frequency with rectal blood loss for which UC therapy was intensified) in their medical history.
6. Subjects who have relapsed on maintenance therapy after 2 weeks with doses of mesalamine at: a. <2.0g/day, will be allowed into the Acute Phase at 2.4g/day QD, or b. between 2.0g/day - 3.0g/day will be allowed into the Acute Phase at 4.8g/day QD.

Inclusion Criteria - Maintenance Phase:

1. Subjects determined to be quiescent at study entry on prior oral mesalamine therapy will be eligible to enter directly into the Maintenance Phase.
2. UC must have been considered to be quiescent, with scores of zero for both rectal bleeding and bowel movements.

Exclusion Criteria - Acute Phase:

1. Subjects who have been in relapse for >6 weeks.
2. Female subjects who are pregnant or lactating, including females with a positive pregnancy test at screening.
3. Subjects must not have used another investigational agent within the last 30 days prior to enrollment.
4. Subjects who have unsuccessfully treated their current relapse with steroids or a mesalamine dose of >2.0 g/day.
5. Subjects who have relapsed on maintenance therapy with doses of mesalamine >2.0g/day. If the subject had a recent dose reduction from 2.0g/day to less than or equal to 2.0g/day and relapsed within 2 weeks of that dose reduction, the subject will not be eligible.
6. Subjects who have used systemic or rectal steroids within the last 4 weeks prior to Baseline, immunosuppressants within the last 6 weeks, antibiotic use within the last 7 days or chronic use of any anti-inflammatory drugs within 7 days prior to Baseline.
7. Subjects with hypersensitivity to salicylates/aspirin are excluded.
8. Subjects with moderate or severe hepatic impairment.
9. Subjects with Crohn's Disease, proctitis (where the extent of inflammation is less than or equal to 15cm), short bowel syndrome, bleeding disorders, or active peptic ulcer disease.
10. Subjects with asthma are excluded only if they are known to be mesalamine-sensitive.
11. Subjects with a positive stool culture for enteric pathogens (including Salmonella, Shigella, Yersinia, Aeromonas, Plesiomonas or Campylobacter) are excluded, as are those with C. difficile toxin present or with ova or parasites as detected by microscopy.
12. Subjects who have a history of previous colonic surgery.
13. Subjects with moderate or severe renal impairment are contra-indicated for treatment with mesalamine compounds and are excluded from the study.
14. Subjects with current or recurrent disease that could affect the colon, the action, absorption or disposition of the study drug, or clinical or laboratory assessments.
15. Subjects with current or relevant previous history of serious, severe or unstable (acute or progressive) physical or psychiatric illness, any medical disorder that may require treatment or make the patient unlikely to fully complete the study, or any condition that presents undue risk from the study drug or procedures.
16. Subjects with a history of alcohol or other substance abuse within the previous year.
17. Subjects who withdrew from a mesalamine trial due to a possibly or probably related severe AE or SAE are not eligible to enter this study.

Exclusion Criteria - Maintenance Phase (in addition to above inclusion for the Acute Phase):

1. Subjects who have withdrawn from the Acute Phase before study visit A3.
2. Subjects with severe UC according to the PGA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2007-05-01 (Actual); Primary Completion 2009-08-17 (Actual); Study Completion 2009-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (62):
- United States (62):
  - Birmingham Gastroenterology Assoc., Birmingham, Alabama
  - Clopton Clinic, Jonesboro, Arkansas
  - VA Medical Center - Long Beach, Long Beach, California
  - Sharp Rees-Stealy Medical Group, San Diego, California
  - Clinical Applications Laboratories, Inc., San Diego, California
  - South Denver Gastroenterology, P.C., Englewood, Colorado
  - The Center for GI Medicine of Fairfield & Westchester, P.C., Greenwich, Connecticut
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Connecticut Gastroenterology Associates, New Haven, Connecticut
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Advanced Digestive Care, PA, Clearwater, Florida
  - Southern Clinical Research Consultants, Hollywood, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - United Medical Research, New Smyrna Beach, Florida
  - Advanced Gastroenterology Associates, Palm Harbor, Florida
  - Soapstone Ctr. for Clin. Rsrch, Decatur, Georgia
  - Gastroenterology Assoc./Cen.GA, Macon, Georgia
  - NW GA Gastroenterology, Marietta, Georgia
  - Midwest Clinical Research Associates, Moline, Illinois
  - Accelovance, Peoria, Illinois
  - Rockford Gastroenterology Associates, Rockford, Illinois
  - Indiana University Hospital, Indianapolis, Indiana
  - Gastrointestinal Clinic of Quad Cities, Davenport, Iowa
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - GI Associates, Overland Park, Kansas
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Digestive Disorders Associates Research Division, Annapolis, Maryland
  - Maryland Clinical Trials, Annapolis, Maryland
  - Maryland Digestive Disease Research, LLC, Laurel, Maryland
  - Center for Digestive Health, Troy, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Center for Digestive and Liver Diseases, Mexico, Missouri
  - Clinical Research Group of Montana, PLLC, Bozeman, Montana
  - Marlboro Gastroenterology, Manalapan, New Jersey
  - Western Suffolk Gastroenterology Associates, LLP, Bay Shore, New York
  - Long Island Clinical Research Associates, LLP, Long Island City, New York
  - North Shore University Hospital, Manhasset, New York
  - Winthrop University Hospital, Mineola, New York
  - Digestive Medicine of Long Island, New Hyde Park, New York
  - Mount Sinai and Metropolitan Hospital, New York, New York
  - Upstate Gastroentrology Associates, Troy, New York
  - Peters Medical Research, High Point, North Carolina
  - East Carolina Gastroenterology, Jacksonville, North Carolina
  - Gastroenterology Associates, Beachwood, Ohio
  - Consultants for Clinical Research, Inc., Cincinnati, Ohio
  - Digestive Health Network, Cincinnati, Ohio
  - Gastro Consultants of Greater Cincinnati, Cincinnati, Ohio
  - Gild Consultants, P.C., Dayton, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - Guthrie Clinic, Sayre, Pennsylvania
  - ClinSearch, Chattanooga, Tennessee
  - Gastroenterology of Midsouth, Germantown, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Houston Endoscopy & Research Center, Houston, Texas
  - Gastroenterology Clinic of San Antonio, San Antonio, Texas
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - New River Valley Research, Christiansburg, Virginia
  - Inland Empire Gastroenterology, P.S., Spokane, Washington
  - Spokane Digestive Disease Center, P.S., Spokane, Washington
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Aurora Health Center- Waukesha, Waukesha, Wisconsin

REFERENCES:
- [Result] Kane S, Katz S, Jamal MM, Safdi M, Dolin B, Solomon D, Palmen M, Barrett K. Strategies in maintenance for patients receiving long-term therapy (SIMPLE): a study of MMX mesalamine for the long-term maintenance of quiescent ulcerative colitis. Inflamm Bowel Dis. 2012 Jun;18(6):1026-33. doi: 10.1002/ibd.21841. Epub 2011 Aug 11. PMID 21837775
- [Derived] Yarlas A, Yen L, Hodgkins P. The relationship among multiple patient-reported outcomes measures for patients with ulcerative colitis receiving treatment with MMX (R) formulated delayed-release mesalamine. Qual Life Res. 2015 Mar;24(3):671-83. doi: 10.1007/s11136-014-0797-2. Epub 2014 Sep 6. PMID 25193617
- See also: FDA recall information — http://www.fda.gov/opacom/7alerts.html
- See also: FDA-approved label — http://www.lialda.com/Professional/pdf/pi.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 290 subjects were enrolled in the study (138 in the acute phase and 152 that went directly into the maintenance phase). The 56 subjects that completed the acute phase entered the maintenance phase making a total of 208 subjects in the maintenance phase of the study.
Groups:
- Multi-Matrix System (MMX) Mesalamine: Subjects whose ulcerative colitis (UC) was in flare at screening were enrolled in the 2-month acute phase (MMX Mesalamine dosed orally once-daily [QD] at 2.4-4.8 g/day), while those whose ulcerative colitis was quiescent at screening were enrolled directly into the 12-month maintenance phase (MMX Mesalamine dosed orally QD at 2.4 g/day). Subjects who were treated in the acute phase and attained quiescence were continued into the maintenance phase.
Period: Acute Phase
Arm/Group | Multi-Matrix System (MMX) Mesalamine
Started | 138
Completed | 56
Not Completed | 82
Not completed — Lack of Efficacy | 64
Not completed — Protocol Violation | 10
Not completed — Consent withdrawn | 4
Not completed — Lost to Follow-up | 2
Not completed — Physician Decision | 1
Not completed — noncompliance | 1
Period: Maintenance Phase
Arm/Group | Multi-Matrix System (MMX) Mesalamine
Started | 208
Completed | 138
Not Completed | 70
Not completed — Lack of Efficacy | 40
Not completed — Protocol Violation | 7
Not completed — Adverse Event | 6
Not completed — Consent withdrawn | 5
Not completed — Lost to Follow-up | 3
Not completed — Pregnancy | 1
Not completed — noncompliance | 2
Not completed — prohibited medication use | 2
Not completed — antibiotic use | 1
Not completed — study closure | 1
Not completed — hydrocodone use | 1
Not completed — concomitant medication use | 1

BASELINE CHARACTERISTICS:
Groups:
- MMX Mesalamine (Maintenance Phase): Subjects whose ulcerative colitis was quiescent at screening were enrolled directly into the 12-month maintenance phase (MMX Mesalamine dosed orally QD at 2.4 g/day). Subjects who were treated in the acute phase and attained quiescence were continued into the maintenance phase. A total of 208 subjects entered the maintenance phase (152 whose UC was quiescent at screening + 56 whose UC was quiescent after the acute phase).
Arm/Group | MMX Mesalamine (Maintenance Phase)
Number analyzed (Participants) | 208
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 185
  >=65 years | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (13.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108
  Male | 100
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 208

OUTCOME MEASURES:

1. Primary Outcome: Clinical Recurrence of Ulcerative Colitis (UC) During the Maintenance Phase at 6 Months
Description: Clinical recurrence is defined as 4 or more bowel movements per day above the subject's normal frequency and associated with any of the following: urgency, abdominal pain, or rectal bleeding.
Time Frame: 6 months
Population: Maintenance phase efficacy population (MPEP) includes all subjects who, during the maintenance phase, took at least 1 dose of study medication and had at least 1 post-dose efficacy assessment.
Measure: Number; unit: participants
Groups:
- MMX Mesalamine (Maintenance Phase): Subjects whose ulcerative colitis was in flare at screening were enrolled in the 2-month acute phase (MMX Mesalamine dosed QD at 2.4-4.8 g/day), while those whose ulcerative colitis was quiescent at screening were enrolled directly into the 12-month maintenance phase (MMX Mesalamine dosed QD at 2.4 g/day). Subjects who were treated in the acute phase and attained quiescence were continued into the maintenance phase.
Arm/Group | MMX Mesalamine (Maintenance Phase)
Number analyzed (Participants) | 207
participants
  Yes | 46
  No | 150
  Missing | 11

2. Secondary Outcome: Clinical Recurrence of UC During the Maintenance Phase at 12 Months
Description: as for outcome 1
Time Frame: 12 Months
Population: MPEP
Measure: Number; unit: participants
Arm/Group | MMX Mesalamine (Maintenance Phase)
Number analyzed (Participants) | 207
participants
  Yes | 69
  No | 125
  Missing | 13

3. Secondary Outcome: Clinical Recurrence of UC During the Maintenance Phase Associated With Subject Compliance at 6 Months
Description: Clinical recurrence is defined as 4 or more bowel movements per day above the subject's normal frequency and associated with any of the following: urgency, abdominal pain, or rectal bleeding. Compliance is a subject's adherence to a recommended course of treatment and for this study is calculated: [(Sum of days' supplies dispensed) divided by (Sum of days in all refill intervals)] x 100.
Time Frame: 6 Months
Population: MPEP with non-missing data for clinical recurrence at 6 months.
Measure: Number; unit: Percent of participants
Arm/Group | MMX Mesalamine (Maintenance Phase)
Number analyzed (Participants) | 196
Percent of participants
  < 80% Compliant (n = 36) | 36.1
  80-120% Compliant (n = 158) | 20.9
  > 120% Compliant (n = 2) | 0

4. Secondary Outcome: Clinical Recurrence of UC During the Maintenance Phase Associated With Subject Compliance at 12 Months
Description: Clinical recurrence is defined as 4 or more bowel movements per day above the subject's normal frequency and associated with any of the following: urgency, abdominal pain, or rectal bleeding. Compliance is a subject's adherence to a recommended course of treatment and for this study is calculated: (Sum of days' supplies dispensed) divided by (Sum of days in all refill intervals) x 100.
Time Frame: 12 months
Population: MPEP with non-missing data for clinical recurrence at 12 months.
Measure: Number; unit: Percent of participants
Arm/Group | MMX Mesalamine (Maintenance Phase)
Number analyzed (Participants) | 194
Percent of participants
  < 80% Compliant (n = 40) | 52.5
  80-120% Compliant (n = 154) | 31.2

5. Secondary Outcome: Quiescent UC During the Maintenance Phase at 12 Months
Description: Quiescent UC is defined as scores of 0 for both rectal bleeding and bowel movements. Rectal bleeding is assessed on a scale from 0-3 (0 = no rectal bleeding, 1 = streaks of blood, 2 = obvious blood, 3 = mostly blood). Bowel movements are assessed on a scale of 0-2 (0 = 0-1 more than normal per day, 1 = 2-3 more than normal per day, 2 = 4 or more than normal per day).
Time Frame: 12 Months
Population: MPEP with non-missing data at 12 months.
Measure: Number; unit: Participants
Arm/Group | MMX Mesalamine (Maintenance Phase)
Number analyzed (Participants) | 126
Participants | 101

6. Secondary Outcome: Endoscopic Remission of UC During the Maintenance Phase at 12 Months
Description: Endoscopic remission is defined as an endoscopy score of less than or equal to 1. Endoscopy score (mucosal appearance) ranges from 0-3 (0 = normal [intact vascular pattern; no friability or granulation], 1 = mild [erythema; decreased vascular pattern; minimal granularity], 2 = moderate [marked erythema; granularity; friability; absent vascular pattern; bleeding with minimal trauma; no ulcerations], 3 = severe [ulceration; spontaneous bleeding].
Time Frame: 12 Months
Population: MPEP with non-missing data at 12 months.
Measure: Number; unit: Participants
Arm/Group | MMX Mesalamine (Maintenance Phase)
Number analyzed (Participants) | 132
Participants | 124

ADVERSE EVENTS:
Description: Safety population defined as all subjects who took at least one dose of study medication. In the acute phase 138 were randomized, but only 137 received at least one dose of study medication.
Groups:
- MMX Mesalamine (Acute Phase): Subjects whose ulcerative colitis was in flare at screening were enrolled in the 2-month acute phase (MMX Mesalamine dosed QD at 2.4-4.8 g/day).
- MMX Mesalamine (Maintenance Phase): Subjects whose ulcerative colitis was quiescent at screening were enrolled directly into the 12-month maintenance phase (MMX Mesalamine dosed QD at 2.4 g/day). Subjects who were treated in the acute phase and attained quiescence were continued into the maintenance phase.
Arm/Group | MMX Mesalamine (Acute Phase) | MMX Mesalamine (Maintenance Phase)
Serious Adverse Events (participants affected / at risk) | 3/137 | 9/208
Other Adverse Events (participants affected / at risk) | 0/137 | 12/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MMX Mesalamine (Acute Phase) (N=137) | MMX Mesalamine (Maintenance Phase) (N=208)
Atrial fibrilation (Cardiac disorders) | 1 | 0
Stent occlusion (Injury, poisoning and procedural complications) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Hematochezia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MMX Mesalamine (Acute Phase) (N=137) | MMX Mesalamine (Maintenance Phase) (N=208)
Sinusitis (Infections and infestations) | 0 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.